CLINICAL TRIAL: NCT06446232
Title: Influenza Vaccine Effectiveness in Inpatient and Outpatient Settings Among Young Children in Taiwan
Brief Title: Influenza Vaccine Effectiveness in Among Young Children in Taiwan
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202304120RINC
Record Dates: First submitted 2023-06-27; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Influenza Vaccine Allergy
Keywords: Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project uses questionnaires to statistically analyze whether influenza vaccination is protective for young children.

DETAILED DESCRIPTION:
This plan is expected to admit 350 children who are admitted to the emergency department or hospitalized due to influenza and are aged from 6 months (inclusive) to under 18 years old. Vaccine status, statistical analysis of whether the flu vaccine is protective.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of influenza by Flu A+B rapid antigen test
* Known vaccination status

Exclusion Criteria:

* Unknown vaccination status

Ages: 6 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Those who have performed a rapid influenza screening test, regardless of whether the result is negative or positive
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaires | 12 months
  This project uses questionnaires to statistically analyze whether the flu vaccine is protective for young children. Researchers collect flu rapid test results and invite subjects to write questionnaires. Data collectors administered a standardised questionnaire that included information on demographics, medical history (including flu vaccination status and self-reported prior flu infection).

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan